CLINICAL TRIAL: NCT05382793
Title: Assessment of the Daily Average Requirement of Iodine in Lactating Women: A Dose-response Metabolic Balance Study
Brief Title: Assessment of the Daily Average Requirement of Iodine in Lactating Women
Acronym: LISA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: ETH Zurich (Switzerland) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BASEC2022-00130
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy; Iodine Deficiency
Keywords: Iodine; Dietary requirement; Lactating women; Infant
MeSH Terms: interventions — Iodides; Iodine

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, controlled, dose-response metabolic balance study with cross-over design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactating women with assumed adequate habitual iodine intake (Experimental): Women who consumed iodine-containing dietary supplements during pregnancy (≥150 μg/day). Women in this group will receive a daily oral iodine supplement providing 150 μg iodine as potassium iodide for 14 days before the study start.
  Interventions: Dietary Supplement: Control; Dietary Supplement: Iodide (150 μg/day); Dietary Supplement: Iodine (300 μg/day)
- Lactating mothers with assumed inadequate habitual iodine intake (Experimental): Women who did not consume iodine-containing dietary supplements during pregnancy (≥150 μg/day).
  Interventions: Dietary Supplement: Control; Dietary Supplement: Iodide (150 μg/day); Dietary Supplement: Iodine (300 μg/day)

INTERVENTIONS:
Dietary Supplement: Control — No iodine
Dietary Supplement: Iodide (150 μg/day) — A single oral tablet once daily for five days providing 150 μg iodine as potassium iodide
  Other Names: Jodetten® 150 Henning, Sanofi-Aventis Germany GmbH, Germany
Dietary Supplement: Iodine (300 μg/day) — Two oral tablets (150 μg + 150 μg) daily for five days providing 300 μg iodine as potassium iodide
  Other Names: Jodetten® 150 Henning, Sanofi-Aventis Germany GmbH, Germany

SUMMARY:
Human milk is the only source of iodine during early infancy and adequate iodine intake during lactation is necessary to assure optimal thyroid function in breastfed infants. However, the physiological requirement of iodine in lactating women is uncertain and recommendations for the daily dietary average requirement are poorly defined. WHO recommends iodine supplementation to lactating women in populations with incomplete coverage of iodized salt and deficient iodine intake, but the scientific evidence is weak and the optimal dose is uncertain.

The primary objective is to assess the daily dietary average requirement for iodine in lactating women.

Secondary objectives are to:

* Estimate the daily average requirement for iodine in exclusively breastfed infants;
* Assess the dose-response of dietary iodine supplements on breast milk iodine concentration in lactating women with adequate and inadequate habitual iodine intakes;
* Estimate the maternal iodine intake required to provide exclusively breastfed infants with an adequate iodine intake via breast milk.

DETAILED DESCRIPTION:
This study is a single center, randomized, controlled, dose-response metabolic balance study with cross-over design. The study will be conducted in 24 exclusively breastfeeding women and their infants receding in Zürich, Switzerland. The study involves an initial screening, a 2 weeks run-in period and a balance period over 3 weeks. Participating women will be allocated to two groups based on their consumption of dietary iodine supplements during pregnancy. Women who consumed daily iodine supplements during pregnancy will be assigned to group 1 (n=12) and receive daily supplements containing 150 µg iodine for 2 weeks, whereas women who did not will be enrolled in group 2 and will receive no supplement during the run-in period. Breast milk and spot urine samples (mothers and infants) will be collected daily in all participants during two weeks for the measurement of breast milk and urinary iodine concentrations. During the balance period, all women will receive either no supplement, iodine supplements providing 150 µg/day, or 300 µg/day in random order with cross-over design. Each supplement dose will be assessed in a test period of 7 days, including 2 run-in days, 3 balance days and 2 wash-out days. The supplements will be consumed during the first 5 days in each test-period. During the 3 balance days, the daily iodine intake and excretion will be measured in mothers and infants, and the iodine retention will be calculated for each regimen and study group. The minimum daily average requirement will be determined as the iodine intake where the iodine retention is zero.

ELIGIBILITY:
Mother-infant pairs in good health, free of any acute illness or chronic thyroid disease.

Mothers

Inclusion criteria:

1. Consent to enroll herself and her baby;
2. Age 18 to 49 years;
3. Singleton pregnancy;
4. Exclusively breastfeeding;
5. Self-estimated BMI <30 kg/m2 before conception.

Exclusion criteria:

1. TSH >6 mIU/L;
2. Anemia (Hb <11.7 g/L);
3. Pregnancy (self-reported);
4. Acute illness (e.g. gastroenteritis);
5. History of thyroid disease, diabetes, metabolic disease or inflammatory bowel disease (self-reported);
6. Currently smoking (>1 cigarette/day);
7. Drug abuse or extensive alcohol intake;
8. Exposure to iodine-containing X-ray or computed tomography contrast agents during the past 6 months;
9. Adenomatous goiter, dermatitis, anti-C1q-vasculitis.

Infants

Inclusion criteria:

1. Full term (38-42 weeks);
2. Birthweight ≥2.5 kg;
3. Exclusively breastfed;
4. Age 0-10 weeks at recruitment.

Exclusion criteria:

1. Age >6 months;
2. TSH >10 mIU/L at neonatal screening at 2-5 days after birth (i.e. infants not requested to attend recall assessment);
3. Diagnosed or suspected colic.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 17 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Maternal iodine retention (μg/day) | 24 hours
  Calculated as iodine intake (µg/day) minus the iodine excretion (µg/day)

SECONDARY OUTCOMES:
Maternal iodine excretion in breast milk (μg/day) | 24 hours
  Estimated from measured breast milk iodine concentration (μg/L) and breast milk volume (L)
Infant iodine retention (μg/day) | 24 hours
  Calculated as iodine intake (µg/day) minus the iodine excretion (µg/day)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Braegger, M.D., Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- Nutrition Research Unit, University Children's Hospital Zurich, Zurich, Switzerland